CLINICAL TRIAL: NCT04185883
Title: A Phase 1b, Protocol Evaluating the Safety, Tolerability, Pharmacokinetics, and Efficacy of Sotorasib Monotherapy and in Combination With Other Anti-cancer Therapies in Subjects With Advanced Solid Tumors With KRAS p.G12C Mutation (CodeBreak 101)
Brief Title: Sotorasib Activity in Subjects With Advanced Solid Tumors With KRAS p.G12C Mutation (CodeBreak 101)
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 20190135; 2023-506794-35 (Other: CTIS)
Expanded Access: NCT04667234 (No longer available)
Record Dates: First submitted 2019-12-03; First posted 2019-12-04 (Actual); Last update posted 2025-10-22 (Actual); Status verified 2025-10

CONDITIONS: Advanced Solid Tumors; Kirsten Rat Sarcoma (KRAS) pG12C Mutation
MeSH Terms: interventions — sotorasib; trametinib; Afatinib; pembrolizumab; Panitumumab; Carboplatin; Pemetrexed; Docetaxel; Paclitaxel; atezolizumab; palbociclib; Bevacizumab; Drug Therapy; Everolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (14):
- Sotorasib + trametinib + panitumumab (Experimental): Experimental: Sotorasib + trametinib + panitumumab Dose Exploration and Dose Expansion
  * Enrollment into the dose exploration cohort is for eligible participants with KRAS P.G12C mutant advanced solid tumors.
  * Upon completing the dose exploration part of the study, dose expansion may proceed consisting of participants with KRAS p.G12C mutant advanced solid tumors.
  Interventions: Drug: Sotorasib; Drug: Trametinib; Drug: Panitumumab
- Sotorasib + RMC-4630 (Experimental): Experimental: Sotorasib + RMC-4630 Dose Exploration and Dose Expansion
  * Enrollment into the dose exploration cohort is for eligible participants with KRAS P.G12C mutant advanced solid tumors.
  * Upon completing the dose exploration part of the study, dose expansion may proceed consisting of participants, with KRAS p.G12C mutant advanced solid tumors.
  Interventions: Drug: Sotorasib; Drug: RMC-4630
- Sotorasib + afatinib (Experimental): Experimental: Sotorasib + afatinib Dose Exploration and Dose Expansion
  * Enrollment into the dose exploration cohort is for eligible participants with KRAS P.G12C advanced non-small cell lung cancer.
  * Upon completing the dose exploration part of the study, dose expansion may proceed consisting of participants with KRAS p.G12C mutant advanced non-small cell lung cancer.
  Interventions: Drug: Sotorasib; Drug: Afatinib
- Sotorasib + panitumumab +/- chemotherapy (Experimental): Experimental: Sotorasib + panitumumab +/- chemotherapy Dose Exploration and Dose Expansion
  * Enrollment into the dose exploration cohort is for eligible participants with KRAS P.G12C mutant advanced colorectal cancer.
  * Upon completing the dose exploration part of the study, dose expansion may proceed consisting of participants with KRAS p.G12C mutant advanced solid tumors.
  Interventions: Drug: Sotorasib; Drug: Panitumumab; Drug: IV Chemotherapy (Regimen 1)
- Sotorasib + atezolizumab (Experimental): Experimental: Sotorasib + atezolizumab Dose Exploration and Dose Expansion
  * Enrollment into the dose exploration cohort is for eligible participants with KRAS P.G12C advanced non-small cell lung cancer.
  * Upon completing the dose exploration part of the study, dose expansion may proceed consisting of participants with KRAS p.G12C mutant advanced non-small cell lung cancer.
  Interventions: Drug: Sotorasib; Drug: Atezolizumab
- Sotorasib + carboplatin, pemetrexed, docetaxel, paclitaxel, pembrolizumab (Experimental): Experimental: Sotorasib + carboplatin, pemetrexed, docetaxel, paclitaxel, pembrolizumab Dose Exploration and Dose Expansion
  * Enrollment into the dose exploration cohort is for eligible participants with KRAS P.G12C advanced non-small cell lung cancer.
  * Upon completing the dose exploration part of the study, dose expansion may proceed consisting of participants with KRAS p.G12C mutant advanced non-small cell lung cancer.
  Interventions: Drug: Sotorasib; Drug: Pembrolizumab; Drug: Carboplatin, pemetrexed, docetaxel, paclitaxel
- Sotorasib Monotherapy (Experimental): Experimental: Sotorasib only Dose Exploration and Dose Expansion
  * Enrollment into the dose exploration cohort is for eligible participants with KRAS P.G12C advanced non-small cell lung cancer with brain metastases.
  * Upon completing the dose exploration part of the study, dose expansion may proceed consisting of participants with KRAS p.G12C mutant advanced non-small cell lung cancer with brain metastases.
  Interventions: Drug: Sotorasib
- Sotorasib + palbociclib (Experimental): Experimental: Sotorasib + palbociclib Dose Exploration and Dose Expansion
  * Enrollment into the dose exploration cohort is for eligible participants with KRAS P.G12C advanced solid tumor.
  * Upon completing the dose exploration part of the study, dose expansion may proceed consisting of participants with KRAS p.G12C mutant advanced solid tumor.
  Interventions: Drug: Sotorasib; Drug: Palbociclib
- Sotorasib + pembrolizumab (Experimental): Experimental: Sotorasib + pembrolizumab Dose Exploration and Dose Expansion
  * Enrollment into the dose exploration cohort is for eligible participants with KRAS P.G12C mutant non small cell lung cancer.
  * Upon completing the dose exploration part of the study, dose expansion may proceed consisting of participants with KRAS P.G12C mutant non small cell lung cancer.
  Interventions: Drug: Sotorasib; Drug: Pembrolizumab
- Sotorasib + MVASI® (bevacizumab-awwb)+ Chemotherapy (Experimental): Experimental: Sotorasib + MVASI® (bevacizumab-awwb)+ chemotherapy Dose Exploration and Dose Expansion
  * Enrollment into the dose exploration cohort is for eligible participants with KRAS P.G12C mutant advanced colorectal cancer.
  * Upon completing the dose exploration part of the study, dose expansion may proceed consisting of participants with KRAS p.G12C mutant advanced colorectal cancer.
  Interventions: Drug: Sotorasib; Drug: MVASI® (bevacizumab-awwb); Drug: IV Chemotherapy (Regimen 1); Drug: IV Chemotherapy (Regimen 2)
- Sotorasib + TNO155 (Experimental): Experimental: Sotorasib + TNO155 Dose Exploration and Dose Expansion
  * Enrollment into the dose exploration cohort is for eligible participants with KRAS P.G12C mutant advanced solid tumors.
  * Upon completing the dose exploration part of the study, dose expansion may proceed consisting of participants with KRAS p.G12C mutant advanced solid tumors.
  Interventions: Drug: Sotorasib; Drug: TNO155
- Sotorasib + BI 1701963 (Experimental): Experimental: Sotorasib + BI 1701963 Dose Exploration and Dose Expansion
  * Enrollment into the dose exploration cohort is for eligible participants with KRAS P.G12C mutant advanced solid tumors.
  * Upon completion of dose exploration part of the study the dose expansion cohort is for eligible participants with KRAS P.G12C mutant advanced non-small cell lung cancer and advanced colorectal cancer.
  Interventions: Drug: Sotorasib; Drug: BI 1701963
- Sotorasib + AMG 404 (Experimental): Experimental: Sotorasib + AMG 404 Dose Exploration and Dose Expansion • Enrollment into the dose exploration cohort is for eligible participants with KRAS P.G12C mutant advanced solid tumors. • Upon completing the dose exploration part of the study, dose expansion may proceed consisting of participants with KRAS p.G12C mutant advanced solid tumors
  Interventions: Drug: Sotorasib; Drug: AMG 404
- Sotorasib + everolimus (Experimental): Experimental: Sotorasib + everolimus Dose Exploration and Dose Expansion • Enrollment into the dose exploration cohort is for eligible participants with KRAS P.G12C advanced solid tumor. • Upon completing the dose exploration part of the study, dose expansion may proceed consisting of participants with KRAS p.G12C mutant advanced solid tumor.
  Interventions: Drug: Sotorasib; Drug: Everolimus

INTERVENTIONS:
Drug: Sotorasib — Sotorasib administered orally as a tablet.
Drug: Trametinib — Trametinib administered orally as a tablet.
  Arms: Sotorasib + trametinib + panitumumab
Drug: RMC-4630 — RMC-4630 administered orally as a capsule.
  Arms: Sotorasib + RMC-4630
Drug: Afatinib — afatinib administered orally as a tablet.
  Arms: Sotorasib + afatinib
Drug: Pembrolizumab — pembrolizumab administered as an intravenous (IV) infusion.
  Arms: Sotorasib + carboplatin, pemetrexed, docetaxel, paclitaxel, pembrolizumab; Sotorasib + pembrolizumab
Drug: Panitumumab — Panitumumab administered as an IV infusion.
  Arms: Sotorasib + panitumumab +/- chemotherapy; Sotorasib + trametinib + panitumumab
Drug: Carboplatin, pemetrexed, docetaxel, paclitaxel — Carboplatin, pemetrexed, docetaxel administered as an IV infusion.
  Arms: Sotorasib + carboplatin, pemetrexed, docetaxel, paclitaxel, pembrolizumab
Drug: Atezolizumab — Atezolizumab administered as an IV injection.
  Arms: Sotorasib + atezolizumab
Drug: Palbociclib — Palbociclib administered orally as a tablet.
  Arms: Sotorasib + palbociclib
Drug: MVASI® (bevacizumab-awwb) — MVASI® (bevacizumab-awwb) administered as an IV infusion.
  Arms: Sotorasib + MVASI® (bevacizumab-awwb)+ Chemotherapy
Drug: TNO155 — TNO155 administered orally as a capsule.
  Arms: Sotorasib + TNO155
Drug: IV Chemotherapy (Regimen 1) — Chemotherapy combination of leucovorin administered as an IV injection, 5-fluorouracil (5-FU) administered as IV bolus injection or IV continuous infusion (depending on dose), and irinotecan administered as IV injection.
  Arms: Sotorasib + MVASI® (bevacizumab-awwb)+ Chemotherapy; Sotorasib + panitumumab +/- chemotherapy
Drug: IV Chemotherapy (Regimen 2) — IV chemotherapy combination of leucovorin administered as an IV injection, 5-FU administered as IV bolus injection or IV continuous infusion (depending on dose), and oxaliplatin administered as IV injection.
  Arms: Sotorasib + MVASI® (bevacizumab-awwb)+ Chemotherapy
Drug: BI 1701963 — BI 1701963 administered orally
  Arms: Sotorasib + BI 1701963
Drug: AMG 404 — AMG 404 administered as an IV infusion.
  Arms: Sotorasib + AMG 404
Drug: Everolimus — Everolimus administered orally.
  Arms: Sotorasib + everolimus

SUMMARY:
To evaluate the safety and tolerability of sotorasib administered in investigational regimens in adult participants with KRAS p.G12C mutant advanced solid tumors.

ELIGIBILITY:
Inclusion Criteria:

* Men or women greater than or equal to 18 years old.
* Pathologically documented, locally-advanced or metastatic malignancy with, KRAS p.G12C mutation identified through molecular testing performed according to in-country requirements. In the United States, this test must be performed in a Clinical Laboratory Improvement Amendments (CLIA)-certified laboratory.

Exclusion Criteria:

* Primary brain tumor.
* Spinal cord compression, or untreated, or symptomatic, or active brain metastases, or leptomeningeal disease from non-brain tumors.
* Myocardial infarction within 6 months of study day 1.
* Gastrointestinal (GI) tract disease causing the inability to take oral medication.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 610 (Actual)
Dates: Start 2019-12-17 (Actual); Primary Completion 2026-12-17 (Estimated); Study Completion 2027-12-05 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Dose Limiting Toxicities (DLTs) | 12 Months
Number of Participants with Treatment-emergent Adverse Events (TEAEs) | 12 Months
Number of Participants with Treatment-related Adverse Events | 12 Months
Number of Participants with Clinically Significant Changes in Vital Signs | 12 Months
Number of Participants with Clinically Significant Changes in ECG Measurements | 12 Months
Number of Participants with Clinically Significant Changes in Laboratory Test Values | 12 Months

SECONDARY OUTCOMES:
Maximum Plasma Concentration (Cmax) | 12 Months
Time to Maximum Plasma Concentration (Tmax) | 12 Months
Area Under the Plasma Concentration-time Curve (AUC) | 12 Months
Objective Response Rate | 12 Months
Disease Control Rate | 12 Months
Duration of Response | 12 Months
Progression-free Survival | 12 Months
Duration of Stable Disease | 12 Months
Time to Response | 12 Months
Overall Survival | 12 Months
Sotorasib + EGFR Inhibitor +/- Chemotherapeutic Regimen Only: Quantification of Plasma Levels | 12 Months
Sotorasib Monotherapy Only: Intracranial Objective Response Rate | 12 Months
  Intracranial objective response rate assessed per Response Assessment in Neuro-oncology Brain Metastases (RANO-BM).
Sotorasib Monotherapy Only: Intracranial Disease Control Rate | 12 Months
  Intracranial disease control rate assessed per RANO-BM.
Sotorasib Monotherapy Only: Intracranial Duration of Response | 12 Months
  Intracranial duration of response assessed per RANO-BM.
Sotorasib Monotherapy Only: Time to Intracranial Radiation Therapy | 12 Months
Sotorasib Monotherapy Only: Intracranial Progression-free Survival (PFS) | 12 Months
  Intracranial PFS assessed per RANO-BM.
Sotorasib Monotherapy Only: Non-intracranial Progression-free Survival (PFS) | 12 Months
  Non-intracranial PFS assessed per Response Evaluation Criteria in Solid Tumors (RECIST) 1.1.
Sotorasib Monotherapy Only: Overall Progression-free Survival (PFS) | 12 Months
  Overall PFS assessed per RECIST 1.1 and RANO-BM.
Sotorasib + TNO155 Only: Best Overall Response | 12 Months
Sotorasib + Afatinib + Loperamide Only: Number of Participants with Dose Limiting Toxicities (DLTs) | 12 Months
Sotorasib + Afatinib + Loperamide Only: Number of Participants with Treatment-emergent Adverse Events (TEAEs) | 12 Months
Sotorasib + Afatinib + Loperamide Only: Number of Participants with Treatment-related Adverse Events | 12 Months
Sotorasib + Afatinib + Loperamide Only: Number of Participants with Clinically Significant Changes in Vital Signs | 12 Months
Sotorasib + Afatinib + Loperamide Only: Number of Participants with Clinically Significant Changes in ECG Measurements | 12 Months
Sotorasib + Afatinib + Loperamide Only: Number of Participants with Clinically Significant Changes in Laboratory Test Values | 12 Months

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (90):
- United States (55):
  - Arizona Oncology Associates Professional Corporation, Tucson, Arizona
  - City of Hope National Medical Center, Duarte, California
  - University of California San Diego Moores Cancer Center, La Jolla, California
  - Loma Linda University Cancer Center, Loma Linda, California
  - University of Southern California, Norris Comprehensive Cancer Center, Los Angeles, California
  - University of California Davis Medical Center, Sacramento, California
  - University of California San Francisco Mission Bay Campus, San Francisco, California
  - University of California Los Angeles, Santa Monica, California
  - Rocky Mountain Cancer Centers Denver Midtown, Denver, Colorado
  - Sarah Cannon Research Institute, Denver, Colorado
  - Yale New Haven Hospital, New Haven, Connecticut
  - Norwalk Hospital, Norwalk, Connecticut
  - Memorial Cancer Institute, Pembroke Pines, Florida
  - Moffitt Cancer Center, Tampa, Florida
  - Emory University, Atlanta, Georgia
  - Northwestern University, Chicago, Illinois
  - University of Chicago, Chicago, Illinois
  - Indiana University, Indianapolis, Indiana
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - Johns Hopkins University, Baltimore, Maryland
  - University of Michigan, Ann Arbor, Michigan
  - Henry Ford Cancer Detroit (Brigitte Harris Cancer Pavilion), Detroit, Michigan
  - Washington University, St Louis, Missouri
  - Roswell Park Cancer Institute, Buffalo, New York
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Columbia University Irving Medical Center, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Montefiore Medical Center, The Bronx, New York
  - Levine Cancer Institute, Charlotte, North Carolina
  - Duke University, Durham, North Carolina
  - University of Cincinnati Medical Center, Cincinnati, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Providence Portland Medical Center, Portland, Oregon
  - Oregon Health and Science University, Portland, Oregon
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Gibbs Cancer Center and Research Institute - Spartanburg, Spartanburg, South Carolina
  - Avera Cancer Institute, Sioux Falls, South Dakota
  - United States Oncology Regulatory Affairs Corporate Office, Nashville, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Texas Oncology Central-South, Austin, Texas
  - Mary Crowley Cancer Research, Dallas, Texas
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - Oncology Consultants, Houston, Texas
  - University of Texas MD Anderson Cancer Center, Houston, Texas
  - US Oncology Research Investigational Products Center, The Woodlands, Texas
  - Texas Oncology Northeast Texas, Tyler, Texas
  - Huntsman Cancer Institute, Salt Lake City, Utah
  - University of Virginia Cancer Center, Charlottesville, Virginia
  - Virginia Cancer Specialists, PC, Fairfax, Virginia
  - Fred Hutchinson Cancer Center, Seattle, Washington
  - Northwest Medical Specialties, PLLC, Tacoma, Washington
  - Northwest Cancer Specialists - Vancouver, Vancouver, Washington
- Australia (5):
  - Nepean Cancer Centre, Kingswood, New South Wales
  - GenesisCare -North Shore Oncology, St Leonards, New South Wales
  - Icon Cancer Care South Brisbane, South Brisbane, Queensland
  - The Queen Elizabeth Hospital, Woodville South, South Australia
  - St John of God Healthcare, Subiaco, Western Australia
- Austria (2):
  - Medizinische Universitaet Graz, Graz
  - Landeskrankenhaus Salzburg, Salzburg
- Belgium (2):
  - Universite Catholique de Louvain Cliniques Universitaires Saint Luc, Brussels
  - Universitair Ziekenhuis Antwerpen, Edegem
- CHU de Quebec Hopital de l Enfant Jesus, Québec, Quebec, Canada
- Germany (4):
  - Charite Universitaetsmedizin Berlin, Campus Virchow, Berlin
  - Universitatsklinikum Koln, Cologne
  - Universitaetsklinikum Dresden, Dresden
  - Universitaetsklinikum Essen, Essen
- Italy (3):
  - Azienda Socio Sanitaria Territoriale Grande Ospedale Metropolitano Niguarda, Milan
  - Azienda Ospedaliero Universitaria Pisana, Pisa
  - Centro Ricerche Cliniche Di Verona Societa responsabilita limitata, Verona
- Japan (3):
  - Aichi Cancer Center, Nagoya, Aichi-ken
  - National Cancer Center Hospital East, Kashiwa-shi, Chiba
  - The Cancer Institute Hospital of Japanese Foundation for Cancer Research, Koto-ku, Tokyo
- Universitair Medisch Centrum Utrecht, Utrecht, Netherlands
- South Korea (3):
  - Seoul National University Hospital, Seoul
  - The Catholic University of Korea Seoul St Marys Hospital, Seoul
  - Asan Medical Center, Seoul
- Spain (6):
  - Hospital Universitari Vall d Hebron, Barcelona, Catalonia
  - Hospital Clinic i Provincial de Barcelona, Barcelona, Catalonia
  - Institut Catala d Oncologia Hospitalet Hospital Duran i Reynals, L'Hospitalet de Llobregat, Catalonia
  - Hospital Universitario Puerta de Hierro Majadahonda, Majadahonda, Madrid
  - Hospital Universitario Ramon y Cajal, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
- Taiwan (4):
  - National Cheng Kung University Hospital, Tainan
  - National Taiwan University Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei
  - Linkou Chang Gung Memorial Hospital of Chang Gung Medical Foundation, Taoyuan District
- Sarah Cannon Research Institute UK, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual patient data for variables necessary to address the specific research question in an approved data sharing request
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data sharing requests relating to this study will be considered beginning 18 months after the study has ended and either 1) the product and indication (or other new use) have been granted marketing authorization in both the US and Europe or 2) clinical development for the product and/or indication discontinues and the data will not be submitted to regulatory authorities. There is no end date for eligibility to submit a data sharing request for this study.
Access Criteria: Qualified researchers may submit a request containing the research objectives, the Amgen product(s) and Amgen study/studies in scope, endpoints/outcomes of interest statistical analysis plan, data requirements, publication plan, and qualifications of the researcher(s). In general, Amgen does not grant external requests for individual patient data for the purpose of re-evaluating safety and efficacy issues already addressed in the product labelling. Requests are reviewed by a committee of internal advisors, and if not approved, may be further arbitrated by a Data Sharing Independent Review Panel. Upon approval, information necessary to address the research question will be provided under the terms of a data sharing agreement. This may include anonymized individual patient data and/or available supporting documents, containing fragments of analysis code where provided in analysis specifications. Further details are available at the URL below.
URL: http://www.amgen.com/datasharing

REFERENCES:
- [Background] Kuboki Y, Fakih M, Strickler J, Yaeger R, Masuishi T, Kim EJ, Bestvina CM, Kopetz S, Falchook GS, Langer C, Krauss J, Puri S, Cardona P, Chan E, Varrieur T, Mukundan L, Anderson A, Tran Q, Hong DS. Sotorasib with panitumumab in chemotherapy-refractory KRASG12C-mutated colorectal cancer: a phase 1b trial. Nat Med. 2024 Jan;30(1):265-270. doi: 10.1038/s41591-023-02717-6. Epub 2024 Jan 4. PMID 38177853
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com